CLINICAL TRIAL: NCT03453853
Title: The Study for Atrial Functional Mitral Regurgitation Response In Mitral Loop Cerclage Annuloplasty (AFRICA Study): Multi-center, Open Label, Single Arm, Feasibility Test
Brief Title: Atrial Functional Mitral Regurgitation Response In Mitral Loop Cerclage Annuloplasty (AFRICA Study)
Acronym: AFRICA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong-Hyun Park,MD,PhD, Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFRICA
Record Dates: First submitted 2018-02-12; First posted 2018-03-05 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Atrial Functional Mitral Regurgitation; Heart Failure
Keywords: Percutaneous mitral valve repair; Coronary sinus annuloplasty; Mitral loop cerclage; atrial fibrillation; Mitral Regurgitation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitral Loop Cerclage (Experimental): Intervention: Device: Mitral Loop Cerclage Annuloplasty with CSTV Protective Device
  Interventions: Device: Mitral Loop Cerclage Annuloplasty

INTERVENTIONS:
Device: Mitral Loop Cerclage Annuloplasty — Atrial Functional mitral regurgitation Response In mitral loop Cerclage Annuloplasty
  Other Names: (MLC-B-45-75-R and other 11 models)

SUMMARY:
To evaluate second stage safety and feasibility of Mitral Loop Cerclage(MLC) Annuloplasty with CSTV for repair of functional mitral regurgitation.

DETAILED DESCRIPTION:
The objective of this prospective, single-center, open label, feasibility test is to assess the safety and efficacy of Mitral Loop Cerclage Annuloplasty with CSTV protective device, in treating functional mitral regurgitation (FMR) associated with heart failure and Atrial Fibrillation mitral regurgitation Response in Mitral Loop Cerclage annuloplasty.

ELIGIBILITY:
Inclusion Criteria:

* NYHA(New York Heart Association) Class III - IV
* and, Functional Mitral Regurgitation 3+ (Moderate/Severe) or 4+ (Severe) in spite of optimal medical treatment.

(For optimal medical treatments, ①ACE inhibitor or angiotensin receptor blocker ②β-blocker ③ aldosterone antagonists should be given for at least 3 months unless the subject has contraindication for each drug)

* and, Chronic Atrial Fibrillation in electrocardiography (Persistent AF or Permanent AF)

Exclusion Criteria:

* Primary Mitral Regurgitation
* LV ejection fraction lower than 30%
* Pulmonary arterial pressure ≥ 60mmHg
* End-diastolic Left ventricular dimension ≥ 70mm
* Subjects with functional MR who need CABG or AVR performed
* Pre-existing stent in a coronary artery that is deemed to be in direct contact with the path of mitral loop cerclage along coronary sinus
* Subjects who have functional MR caused by aortic valve disease
* Subjects who have uncontrollable hyperthyroidism
* Subjects who have severe TR due to primary valve leaflet disease
* Anomaly of Coronary Sinus
* Pre-existing devices in coronary sinus such as Implantable Cardioverter Defibrillator and Pacemaker
* 2:1 Atriventricular AV block or higher AV block and ventricular tachycardia
* Subjects with primary MR
* Subjects who cannot be screened by cardiac CT
* Subjects who have possibility of coronary artery pinching even with Mitral Loop Cerclage system judged by cardiac CT
* Subjects who do not have septal vein or have unsuitable septal vein anatomy by cardiac CT or venogram
* Subjects who have thrombosis and embolism
* Creatinine ≥2.0 mg/dL
* Subjects who have coagulation disorders
* Subjects who are unable to take anti-platelet agents
* Pre-existing devices such as Implantable Cardioverter Defibrillator and Pacemaker
* Subjects who are pregnant, or lactating, or plan pregnancy during the clinical trials
* Subjects who are participated in other clinical trials within 1 month of enrollment
* Subjects who are deemed not to be eligible in this study by physician's discretion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
Change of mitral regurgitation severity(1) | 1 month
  changing regurgitant volume (RV,mL) compared with baseline
Change of mitral regurgitation severity(2) | 1 month
  changing effective regurgitant orifice (ERO,cm^2) compared with baseline
Change in mitral annulus geometry | 1 month
  septal lateral dimension(mm)
Rate of adverse events as a measure of safety | 1 month
  Rate of composite endpoint of MACE (Major Adverse Cardiac Event) *death, myocardial infarction, cardiac tamponade, device related cardiac surgery, stroke

SECONDARY OUTCOMES:
Change of mitral regurgitation severity(1) | 6 months
  changing regurgitant volume (RV,mL) compared with baseline
Change of mitral regurgitation severity(2) | 6 months
  changing effective regurgitant orifice (ERO,cm^2) compared with baseline
Change in mitral annulus geometry | 6 months
  septal lateral dimension(mm)
Change in left ventricle volumes | 6 months
  Changing of End-diastolic phase LV volumes(mL)
Electrical remodeling | 6 months
  change in electrocardiography (conversion of atrial fibrillation to normal sinus rhythm)
Change in subjects' symptoms referred to NYHA Classification System | 6 months
  NYHA (New York Heart Association)
Technical success rate of the implantation | 6 months
  Technical feasibility by the implantation success rate (%)
Rate of adverse events as a measure of safety | 6 months
  Rate of composite endpoint of MACE (Major Adverse Cardiac Event) *death, myocardial infarction, cardiac tamponade, device related cardiac surgery, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Hyun Park, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (7):
- South Korea (7):
  - Keimyung University Dongsan Hospital, Daegu, Dalseo-gu
  - Sejong HOSPITAL, Bucheon-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chungnam National University Hospital (CNU Hospital), Daejeon, Jung-gu
  - Yeungnam University Hospital, Daegu, Nam-gu
  - Ulsan Hospital, Ulsan, Nam-gu
  - ASAN Medical Center, Seoul, Songpa-gu

REFERENCES:
- [Background] Kim JH, Kocaturk O, Ozturk C, Faranesh AZ, Sonmez M, Sampath S, Saikus CE, Kim AH, Raman VK, Derbyshire JA, Schenke WH, Wright VJ, Berry C, McVeigh ER, Lederman RJ. Mitral cerclage annuloplasty, a novel transcatheter treatment for secondary mitral valve regurgitation: initial results in swine. J Am Coll Cardiol. 2009 Aug 11;54(7):638-51. doi: 10.1016/j.jacc.2009.03.071. PMID 19660696
- [Background] Park YH, Chon MK, Lederman RJ, Sung SC, Je HG, Choo KS, Lee SH, Shin ES, Kim JS, Hwang KW, Lee SY, Chun KJ, Kim CM, Kim JH. Mitral Loop Cerclage Annuloplasty for Secondary Mitral Regurgitation: First Human Results. JACC Cardiovasc Interv. 2017 Mar 27;10(6):597-610. doi: 10.1016/j.jcin.2016.12.282. PMID 28335897